CLINICAL TRIAL: NCT02119975
Title: A Working Memory Training to Decrease Rumination in Depressed and Anxious Individuals: A Double-blind Randomized Controlled Trial
Brief Title: A Working Memory Training to Decrease Rumination in Depressed and Anxious Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ingmar Franken, Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2014-04-08; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Major Depression; Anxiety Disorder
Keywords: Rumination; Working memory; Depression; Anxiety; Working memory training; Overgeneral memories
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Rumination Syndrome; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo working memory training (Placebo Comparator)
  Interventions: Behavioral: Placebo training
- Working memory training (Experimental)
  Interventions: Behavioral: Working memory training

INTERVENTIONS:
Behavioral: Working memory training
  Arms: Working memory training
Behavioral: Placebo training
  Arms: Placebo working memory training

SUMMARY:
Dysfunctioning executive functioning, including working memory (WM), is related to rumination. Findings show that working memory capacity (WMC) can be increased by training. The current study explored by means of a double-blind randomized controlled trial whether an adaptive WM training could reduce rumination, anxiety and depression in a sample of 98 depressed and anxious individuals.

ELIGIBILITY:
Inclusion Criteria:

* Major depression diagnosis
* Anxiety diagnosis

Exclusion Criteria:

* Current psychosis
* Substance abuse

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in Ruminative Response Scale (RRS) score from pre to post training and after two months (follow up 2) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  Dutch version; Raes, Hermans, & Eelen, 2003) measures the frequency of self-reported rumination behavior, with answer options ranging from 1 (never) to 4 (always). The total score of the 22 items was used in the analyses.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory Second Edition (BDI-II) score from pre to post training and after two months (follow up 2) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The Beck Depression Inventory - II (BDI-II; Beck, Steer, & Brown, 1996; Dutch version: Van der Does, 2002) measures the severity of depression symptoms of the last two weeks.
Change in State-Trait Anxiety Inventory (STAI) score from pre to post training and after two months (follow up 2) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The State-Trait Anxiety Inventory (STAI; Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983, Dutch version; Van der Ploeg, Defares, & Spielberger, 1979) measures self-reported anxiety, divided in state anxiety and trait anxiety.

OTHER OUTCOMES:
The change in Internal Shift Task (IST) score from pre to post training and to follow up (two months after post) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The Internal Shift Task (IST; De Lissnyder et al., 2012) measures the ability to shift attention between items stored in WM.
The change in Digit Span score from pre to post training and to follow up (two months after post) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The Digit Span (Lumley & Calhoun, 1934), which consist of two parts: the forward and backward span, with 14 trials each. The forward Digit Span is a frequently used measure for short term memory, an important subcomponent of the memory system (Shipstead et al., 2012) and the backward version measures WM.
The change in Reading Span partial-credit unit score from pre to post training and to follow up (two months after post) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The Reading Span (Daneman & Carpenter, 1980), the third WMC assessment, measures the processing and storage functions of the WM (Shipstead et al., 2012).

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Rotterdam, Rotterdam, South Holland, Netherlands